CLINICAL TRIAL: NCT03347513
Title: Does Eradication of H-pylori in Pregnant Patients With Iron Deficiency Anemia Have an Effect on Iron Replacement Therapy?
Brief Title: Eradication of H-pylori in Pregnancy and Its Effect on Iron Replacement Therapy?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Assistant professor of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A15112017
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy Complications; Anemia, Iron Deficiency; H Pylori Infection
Keywords: H-pylori; iron deficiency anemia; Pregnancy; iron therapy
MeSH Terms: conditions — Pregnancy Complications; Anemia, Iron-Deficiency | interventions — ferroglycine sulfate

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eradication of H-pylori (Experimental): triple attack therapy (Clarithromycin 500 mg BID for 14 days, omeprazole 20 mg BID for 14 days, metronidazole 500 mg BID for 14 days).
  Followed by confirmation of eradication by repeating the H-pylori stool antigen test.
  Iron therapy will be given twice daily for one month in the form ferrous(II)-glycine-sulphate complex 567.7 mg capsules (each capsule contains about 100 mg elemental iron) Ferro sanol duodenal ®Minapharm, Egypt.
  Interventions: Drug: triple attack therapy; Drug: Ferrous(II)-glycine-sulphate complex 567.7 mg capsules
- No eradication of H-pylori (Active Comparator): Iron therapy will be given twice daily for one month in the form ferrous(II)-glycine-sulphate complex 567.7 mg capsules (each capsule contains about 100 mg elemental iron) Ferro sanol duodenal ®Minapharm, Egypt.
  Interventions: Drug: Ferrous(II)-glycine-sulphate complex 567.7 mg capsules

INTERVENTIONS:
Drug: triple attack therapy — eradication of H-pylori using triple attack therapy.
  Other Names: KLACID XL 500 mg; HEALSEC 20 mg; Flagyly 500 mg
  Arms: Eradication of H-pylori
Drug: Ferrous(II)-glycine-sulphate complex 567.7 mg capsules — Iron therapy will be given to both groups twice daily for one month.
  Other Names: Ferro sanol duodenal ®Minapharm , Egypt

SUMMARY:
the effect of eradication of H-pylori in pregnant patients with iron deficiency anemia on the level of hemoglobin after iron therapy.

DETAILED DESCRIPTION:
After approval of the "Ethics Committee" of the obstetrics and gynecology department of the faculty of medicine Cairo University, a clinical trial will be started in which pregnant patients with iron deficiency anemia will be recruited out of the antenatal care clinic. Routine complete blood count (CBC) is done early during the second trimester for cases with anemia discovered by labs drawn on their booking appointment during their 1st antenatal care visit.

IDA defined as hemoglobin below 11gm/dl with MCV below 80 fl, with one of the following: if the serum ferritin level is below 70 μg/L. or if transferrin saturation is below 20.

We based our sample size according to the work done by Nashaat & Mansour, 2014 who studied a difference in the mean hemoglobin level of 1.6 g/dl with a standard deviation of 3.3. The ratio of women in the control group to experimental group was set at 1:1, the power at 0.8, and the type I error at 0.05 which gave us 68 subjects in every arm. We allowed for 10% dropouts finally giving us 75 subjects on each study arm.

After obtaining informed consent, H-pylori infection will be diagnosed using a stool antigen assay ABON which is one step H. pylori antigen test device (®Inverness Medical Innovation Hong Kong Limited). A stool sample will be collected and the top screwed on. An applicator will then be introduced into the sample after unscrewing of the cap in three different sites to collect at least 50 mg of fecal matter. The sample will be centrifuged at 4000 rpm for 5 minutes and the supernatant will be used for immunoassay. Two drops will be placed on the kit as per kit instructions. This test utilizes lateral chromatographic assay where after 10 minutes a positive sample will have a purple-pink line in addition to the control line, while a negative test only has the control line present. If the control line was missing the test will be considered invalid.

All the enrolled participants will then be randomized into two groups using a computer generated randomization table and a sealed envelope system to be opened by the nurse in the next antenatal care visit. When the envelope is opened the participant will be assigned to either group (A) (eradication of H-pylori before iron therapy) or group (B) (start iron therapy without eradication o f H-pylori).

Participants in group A will undergo eradication of H-pylori using triple attack therapy according to O'Connor et al, 2013 with Proton pump inhibitor (eg, omeprazole 20 mg BID), Clarithromycin 500 mg BID, metronidazole 500 mg BID for 14 days, followed by confirmation of eradication by repeating the H-pylori stool antigen test .

Iron therapy will be given to both groups twice daily for one month in the form ferrous(II)-glycine-sulphate complex 567.7 mg capsules (each capsule contains about 100 mg elemental iron) Ferro sanol duodenal ®Minapharm , Egypt. All recruited cases will undergo blood sampling for complete blood count (CBC), serum ferritin, transferrin saturation, and total iron binding capacity (TIBC) before and after iron therapy. All demographic data along with relevant history taking and examination will be recorded at the beginning of recruitment including age, body mass index (BMI), and parity e.t.c.

PS Power and Sample Size Calculations software, version 2.1.30 for MS Windows, was used to calculate sample size (Dupont and Vanderbilt, Nashville, TN).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Iron deficiency anemia.
* H-pylori positive cases.
* Second trimester pregnancy.

Exclusion Criteria:

* Severe Iron deficiency anemia (hemoglobin < 8.0 g/dL).
* Parasitic worm infection e.g. schistosomiasis, and hook worm by stool analysis.
* Any cases giving clinical symptoms of gastritis e.g. nausea, vomiting, dull aching pain or soreness in the epigastrium.
* Cases with history of gastric ulcer diagnosed by upper endoscopy.
* Cases complaining of hematemesis.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
hemoglobin levels | one month
  difference in mean mean hemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamel, M.D., Principal Investigator — Cairo University
Locations (1):
- obstetrics and gynecology department, Kasr Alainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nashaat EH, Mansour GM. Helicobacter pylori and anemia with pregnancy. Arch Gynecol Obstet. 2014 Jun;289(6):1197-202. doi: 10.1007/s00404-013-3138-8. Epub 2013 Dec 28. PMID 24374855
- [Background] Breymann C, Honegger C, Hosli I, Surbek D. Diagnosis and treatment of iron-deficiency anaemia in pregnancy and postpartum. Arch Gynecol Obstet. 2017 Dec;296(6):1229-1234. doi: 10.1007/s00404-017-4526-2. Epub 2017 Sep 22. PMID 28940095
- [Background] Chey WD, Leontiadis GI, Howden CW, Moss SF. ACG Clinical Guideline: Treatment of Helicobacter pylori Infection. Am J Gastroenterol. 2017 Feb;112(2):212-239. doi: 10.1038/ajg.2016.563. Epub 2017 Jan 10. PMID 28071659